CLINICAL TRIAL: NCT02372760
Title: For A More Comfortable Bronchoscopy: Is Spray Catheter The Answer?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has relocated and the study has been closed.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UFJ 2014-47
Record Dates: First submitted 2015-02-03; First posted 2015-02-26 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Airway Complication of Anaesthesia
Keywords: Bronchoscopic anesthesia lidocaine; Spray Catheter; brochoalveolar lavage
MeSH Terms: interventions — Anesthesia; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BA by spray catheter (Olympus PW-205V) (Experimental): This group will be having the bronchoscopic anesthesia (lidocaine) injected through the spray catheter (Olympus PW-205V).
  Interventions: Device: BA by spray catheter (Olympus PW-205V); Drug: Anesthesia
- BA classic anesthesia (Active Comparator): This group will be having the bronchoscopic anesthesia (lidocaine) injected through the bronchoscope's working channel.
  Interventions: Other: BA classic anesthesia; Drug: Anesthesia

INTERVENTIONS:
Device: BA by spray catheter (Olympus PW-205V) — This group will be having the bronchoscopic anesthesia (lidocaine) injected through the spray catheter (Olympus PW-205V)
  Other Names: Spray catheter
  Arms: BA by spray catheter (Olympus PW-205V)
Other: BA classic anesthesia — This group will have the bronchoscopic anesthesia (lidocaine) injected through the bronchoscope's working channel.
  Arms: BA classic anesthesia
Drug: Anesthesia — Both groups will receive lidocaine as the anesthesia for bronchoscopy
  Other Names: Lidocaine

SUMMARY:
Bronchoscopy is a commonly performed procedure for inpatients to visualize the airways when indicated. It is routinely done for both diagnostic (to lavage and biopsy the respiratory tract) and therapeutic purposes (to relief an obstruction or remove foreign bodies). Given the possible side effects of cough of varying severity this procedure can be uncomfortable to patients, some would even shy away from having a bronchoscopy even when it's medically indicated.

Recently a spray catheter was designed to deliver more uniform anesthesia to the airways as compared to the conventional way of injecting the anesthesia into the bronchoscopy working channel. The investigators aim to conduct this study with the hope of improving patient care, providing comfortable procedures, helping more patients opt in for bronchoscopy when indicated.

DETAILED DESCRIPTION:
Bronchoscopy is a commonly performed procedure for inpatients. It is routinely done for both diagnostic and therapeutic purposes. The physician in this procedure inserts the bronchoscopy tube that has a camera at its tip to visualize the airways and detect possible pathologies. When needed, he/she can take samples (biopsies), perform brochoalveolar lavage, remove foreign bodies, or relieve airway obstructions.

The usual method of Bronchoscopic Anesthesia (BA) is conscious sedation combined with local anesthesia as it's more comfortable for the patients, with less chances of lidocaine toxicity. Local anesthesia is classically done using lidocaine injected through the bronchoscope's working channel. As the operator starts from the upper airway, they anesthetize each part as they go down to examine the lungs. The lidocaine will be delivered to the airway as it drips out of the working channel into the airway part closest to it. Side effects of this method is cough with varying frequencies/severity that may sometimes hinder the procedure.

Recently, a spray catheter was designed and used, but mainly for EBUS (Endobronchial Ultrasound) and not for bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age and above)
* Not mechanically ventilated
* Needing a bronchoscopy as determined by a referring or consulting physician/medical service

Exclusion Criteria:

* Individuals below 18 years of age
* Pregnant women
* Terminally-ill patients
* Patients who are unable to consent in person
* Patients with contraindications for bronchoscopy (according to British Thoracic Society 2013 Guidelines this includes patients with acute myocardial infarction and patients in acute respiratory distress)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of coughing episodes during the bronchoscopy | Day 1
  Coughing data will be collected from both groups during the bronchoscopy
Severity of cough during the bronchoscopy | Day 1
  Severity of cough data will be collected from both groups during the bronchoscopy
Endotracheal sedations required to conduct the bronchoscopy | Day 1
  Endotracheal sedations required to conduct the bronchoscopy between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Adil Shujaat, MD, Principal Investigator — University at Buffalo
Locations (1):
- UF Health, Jacksonville, Florida, United States

REFERENCES:
- [Background] Stolz D, Chhajed PN, Leuppi J, Pflimlin E, Tamm M. Nebulized lidocaine for flexible bronchoscopy: a randomized, double-blind, placebo-controlled trial. Chest. 2005 Sep;128(3):1756-60. doi: 10.1378/chest.128.3.1756. PMID 16162784
- [Background] De S. Assessment of patient satisfaction and lidocaine requirement during flexible bronchoscopy without sedation. J Bronchology Interv Pulmonol. 2009 Jul;16(3):176-9. doi: 10.1097/LBR.0b013e3181afca25. PMID 23168547
- [Background] Jakobsen CJ, Ahlburg P, Holdgard HO, Olsen KH, Thomsen A. Comparison of intravenous and topical lidocaine as a suppressant of coughing after bronchoscopy during general anesthesia. Acta Anaesthesiol Scand. 1991 Apr;35(3):238-41. doi: 10.1111/j.1399-6576.1991.tb03280.x. PMID 2038931
- [Background] Antoniades N, Worsnop C. Topical lidocaine through the bronchoscope reduces cough rate during bronchoscopy. Respirology. 2009 Aug;14(6):873-6. doi: 10.1111/j.1440-1843.2009.01587.x. PMID 19703068
- [Background] Lee HJ, Haas AR, Sterman DH, Solly R, Vachani A, Gillespie CT. Pilot randomized study comparing two techniques of airway anaesthesia during curvilinear probe endobronchial ultrasound bronchoscopy (CP-EBUS). Respirology. 2011 Jan;16(1):102-6. doi: 10.1111/j.1440-1843.2010.01861.x. PMID 20920136
- [Background] Kenzaki K, Hirose Y, Tamaki M, Sakiyama S, Kondo K, Mutsuda T, Monden Y. Novel bronchofiberscopic catheter spray device allows effective anesthetic spray and sputum suctioning. Respir Med. 2004 Jul;98(7):606-10. doi: 10.1016/j.rmed.2004.01.002. PMID 15250225
- [Background] Wahidi MM, Jain P, Jantz M, Lee P, Mackensen GB, Barbour SY, Lamb C, Silvestri GA. American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. Chest. 2011 Nov;140(5):1342-1350. doi: 10.1378/chest.10-3361. PMID 22045879
- [Background] Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, Mandal S, Martin J, Mills J, Navani N, Rahman NM, Wrightson JM, Munavvar M; British Thoracic Society Bronchoscopy Guideline Group. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-i44. doi: 10.1136/thoraxjnl-2013-203618. No abstract available. PMID 23860341